CLINICAL TRIAL: NCT06770699
Title: Prognostic Performance of Tertiary Lymphoid Structures in Nasopharyngeal Carcinoma: a Prospective Multi-Center Observational Study
Brief Title: Tertiary Lymphoid Structures in Nasopharyngeal Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TLS-NPC
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinom; Tertiary Lymphoid Structures; Outcome
MeSH Terms: conditions — Tertiary Lymphoid Structures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TLS positive: Positive TLS in Tumor
- TLS negative: no TLS in Tumor

SUMMARY:
This study aims to conduct a prospective cohort study to validate the prognostic performance of Tertiary Lymphoid Structures (TLSs) as a predictive marker in pathological tissue sections for nasopharyngeal carcinoma (NPC). The TLS assessment framework established in this research has the potential to serve as a reference for personalized treatment strategies in NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological confirmed diagnosis of nasopharyngeal carcinoma (NPC).
2. No evidence of distant metastasis at initial treatment, with staging classified as II-III (AJCC 9th edition).
3. Patients aged 18-75 with a Karnofsky Performance Status (KPS) score ≥ 80.
4. Organ Function: Adequate organ function meeting the following criteria:

   * Hematology:

   White blood cell count > 3.0 × 10⁹/L. Absolute neutrophil count (ANC) > 1.5 × 10⁹/L. Hemoglobin (Hb) > 90 g/L. Platelet count > 100 × 10⁹/L. Albumin ≥ 3 g/dL.

   >Liver Function: Bilirubin ≤ 1.5 × the upper limit of normal (ULN); patients with Gilbert's syndrome may enroll if serum bilirubin ≤ 3 × ULN.

   Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN; for patients with liver metastasis, AST/ALT ≤ 5 × ULN.

   Alkaline phosphatase (ALP) ≤ 3 × ULN; for patients with liver or bone metastasis, ALP ≤ 5 × ULN.

   >Coagulation Function: International normalized ratio (INR), prothrombin time (PT), or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

   >Renal Function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 mL/min as calculated by the Cockcroft-Gault formula (see Appendix 8).
5. Patients willing and able to comply with visit schedules, treatment plans, laboratory tests, and other study procedures.
6. Willing to adhere to study arrangements and refrain from participating in any other clinical trials related to drugs or medical devices during the study period.
7. Signed a formal informed consent form, indicating that they understand and agree to participate in the study in compliance with hospital policies.
8. Sufficient tumor tissue stored in paraffin blocks, suitable for scientific research purposes.

Exclusion Criteria:

1. Patients with concurrent malignant tumors other than nasopharyngeal carcinoma.
2. Patients with a history of severe immediate allergic reactions to any drug used in this study.
3. Patients who lack legal capacity or have limited legal capacity.
4. Patients with a history of drug or alcohol abuse, or with physical or mental disorders, who, in the investigator's opinion, are unable to fully understand or comply with the study's procedures and potential complications.
5. Patients with other serious acute or chronic medical conditions, laboratory abnormalities, or mental disorders that may increase the risk of treatment-related adverse events, interfere with the interpretation of study results, or make them unsuitable for participation in the study, as determined by the investigator. These include, but are not limited to:

   Autoimmune colitis, inflammatory bowel disease, noninfectious pneumonitis, pulmonary fibrosis;
6. Mental disorders such as dementia, epilepsy, or recent (within the past year) or active suicidal ideation or behavior.
7. Patients with a prior diagnosis of immunodeficiency or known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related diseases.
8. Pregnant or breastfeeding women, and male or female patients of childbearing potential who are unwilling or unable to use effective contraception throughout the study period and for at least one year after completing the treatment regimen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage II-III Nasopharyngeal Carcinoma
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 3 Years
  DFS is defined as the time from the date of enrollment to the first occurrence of either disease progression (as confirmed by imaging or clinical evaluation) or death from any cause, whichever occurs first. For patients without these events, DFS is censored at the time of the last follow-up.

SECONDARY OUTCOMES:
Overall Survival | 3 Years
  OS is defined as the time from the date of enrollment to death from any cause, or the time interval to the last follow-up for patients who are alive at the end of the study.
Locoregional Recurrenc-free Survival | 3 Years
  LRRFS is defined as the time from the date of enrollment to the first occurrence of locoregional relapse (confirmed by imaging or clinical evaluation), or the time interval to the last follow-up for patients without locoregional relapse.
Distant Metastasis-Free Survival | 3 Years
  DMFS is defined as the time from the date of enrollment to the first occurrence of distant metastasis (confirmed by imaging or clinical evaluation), or the time interval to the last follow-up for patients without distant metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China